CLINICAL TRIAL: NCT04673773
Title: MY RELIEF- Evidence Based Information to Support People Aged 55+ Years Living and Working With Persistent Low-back Pain: Using a Digital Platform
Brief Title: MY RELIEF- Evidence Based Information to Support People Aged 55+ Years Living and Working With Persistent Low-back Pain.
Acronym: MY-RELIEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Collaborators: University of Ulster (Other); Kaunas University of Technology (Other); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Associate Professor, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 018-1-SE01-KA204-039144
Record Dates: First submitted 2020-11-04; First posted 2020-12-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Low Back Pain
Keywords: Low back pain; Older adults; Work
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility / A massive open course (Experimental): 1. The online MOOC contains eight units which cover the following topics (Understanding low back pain (LBP), Physical activity and exercise in relation to LBP, Psychological factors, Sleep / nutrition, Management of LBP at the workplace, Communication with health care, Other issues related to LBP). Each unit will include short factual texts, short videos (2-5mins) with older workers (aged 55+ years) with low back pain and professional experts, as well as knowledge tests. The complete MOOC will take 2-3 hours to complete. It would be possible to complete the MOOC at one time however users will be recommended to complete two units per week over a month period.
  2. The mobile game is designed to encourage participation with the MOOC by providing feedback on engagement with the MOOC, presentation of quizzes to test knowledge gained on the MOOC, as well as feedback on clinical markers of their condition e.g. Mood, pain, physical activity levels.
  Interventions: Behavioral: A Massive Open Online Course

INTERVENTIONS:
Behavioral: A Massive Open Online Course — Same as intervention

SUMMARY:
Low back pain is the main cause of activity limitation and work absence across the world, leading to a high social and economic burden for individuals, families, the labour market and society. This is particularly true for older adults of working age, employed in sedentary or arduous/strenuous jobs, whose work conditions may influence negatively this health problem and lead to severe persistent low back pain. Pain management is one of the most neglected aspects of healthcare and people suffering from persistent low back pain are often left without specific information, guidance and care from healthcare systems.

The MY-RELEF study is a multinational, multicenter, prospective uncontrolled, pre-post intervention feasibility study targeting people over the age of 55 years with persistent low back pain in Northern Lithuania, Ireland, Italy, Sweden and Portugal. Eligible participants will be offered the opportunity to use the MY RELIEF educational platform as part of their care and will undergo evaluations at baseline (enrollment) and at two-weeks and one-month follow-ups.

DETAILED DESCRIPTION:
A Massive Open Online Course (MOOC) called MY RELIEF, have been developed. MY-RELIEF is built on best practices in e-learning, e-health and multimedia-based learning. The training package will be available on mobile devices such as a mobile phone or a tablet. The training is designed in short modules (10-12 minutes per module), possible to complete during a break in work. The MOOC will include short videos with older workers (aged 55+ years) with low back pain and professional experts, as well as knowledge tests and short factual texts. In addition, the target audience will have access to a serious game on their mobile phone that will track their health, and provide feedback on their potentially changing health status, and their engagement with the MOOC units.

The aim for this study is to determinate usability, acceptability and feasibility of a digital education program (MY-RELIEF) delivered via a MOOC for people aged 55+ years with persistent low back pain who are in sedentary or physically demanding jobs, and need advice on ergonomics, self-management of pain and healthy behavioral strategies.

The usability of the intervention will be measured with an industry standard tool to understand peoples ease of interaction with the MOOC and acceptability of the content and format of the MOOC will be measured via qualitative feedback from users.

Feasibility will be informed by the data on likely recruitment and follow up rates in each country for a main trial, floor and ceiling effects and completion rates on outcome measures, and likely within group effect sizes in response to the MOOC.

MY-RELIEF will help to improve and expand the range of high quality learning opportunities tailored to the needs of people over the age of 55 years.

ELIGIBILITY:
Inclusion criteria:

1. Understand Lithuanian (Lithuanian study), English (N Irish study), Italian (Italian study), Swedish (Sweden) and Portuguese (Portugal).
2. Participant is willing and able to give informed consent for participation in the study via the study website.
3. Persistent low back pain; defined as pain between scapulae and gluteal region, with or without radiation towards one or both legs, present for at least three months.
4. Aged over 55 years
5. In employment.

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

1. People with unexplained symptoms
2. People who have not seen a health care professional and received a diagnosis of persistent low back pain
3. People who have been given a diagnosis of specific low back pain
4. People with evidence of serious underlying pathology, such as a current diagnosis of cancer
5. Anyone who has not used or have no interest in using a computer, laptop, tablet or mobile phone.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Retention rates | 4 weeks after baseline
  Of the people who are recruited into the study how many MOOC units do they complete
Recruitment of participants | 4 weeks after baseline
  Percentage of people who participate in the intervention by signing up directly to the website versus the percentage who are recruited via the research team
User satisfaction with the MOOC | 4 weeks after baseline
  Qualitative Semi-structured interviews/focus groups
Usability of the MOOC | 4 weeks after baseline
  System usability Scale(SUS), is a simple, ten-item scale giving a global view of subjective assessments of usability. The selected statements in the SUS are measured on a five point Likert scale and cover a variety of aspects of system usability, such as the need for support, training, and complexity, and thus have a high level of validity for measuring usability of a system. The scale yield a score between 0-100 were high values represent high usability.
Change in Participant's health-related quality of life | At baseline and 4 weeks later
  EQ-5D
Change in Functional disability | At baseline and 4 weeks later
  Functional disability will be measured by the Oswestry Disability Questionnaire. The ODQ consists of 10 sections, each with six levels (with a maximum score in each section of five points) that assess an individual's limitations in various activities of daily living. The sum of all 10 sections is divided by the total possible score and the result multiplied by 100 to generate a percentage score. Values range from 0 (best health state) to 100 (worst health state).
Patient ability to cope with with illness and life after using the MOOC | 4 weeks after baseline
  An adapted version of the Patient enablement Instrument (PEI), a six-item questionnaire designed to measure the patient's ability to understand and cope with illness and life following a consultation with a general practitioner will be used. Given this an adapted version of the PEI will be used, where the words 'after this appointment' and 'as a result of your visit to the doctor today' will be replaced by 'after using the Serious game (MOOC)' and 'as a result of using the Serious game(MOOC)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall-Hansson, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marley J, Larsson C, Piccinini F, Howes S, Casoni E, Hansson EE, McDonough S. Study protocol for a feasibility study of an online educational programme for people working and living with persistent low back pain. Pilot Feasibility Stud. 2023 Sep 4;9(1):154. doi: 10.1186/s40814-023-01382-3. PMID 37667407